CLINICAL TRIAL: NCT06654115
Title: Wireless Vital Sign Monitoring in Women After Cesarean Birth in Pakistan
Brief Title: Wireless Physiologic Monitoring After Cesarean
Acronym: WIP
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Lund University (Other)
Collaborators: Harvard Medical School (HMS and HSDM) (Other); Sir Ganga Ram Hospital (Other); The Swedish Research Council (Other Government)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: LUNDMZ
Record Dates: First submitted 2024-10-21; First posted 2024-10-23 (Actual); Last update posted 2024-10-23 (Actual); Status verified 2024-10

CONDITIONS: Cesarean Section Complications; Vital Signs Monitoring; Maternal Health Care

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- WIP (Active Comparator): wireless biosensor arm
  Interventions: Device: Wireless Physiologic Monitoring
- SOC (No Intervention): Standard of care

INTERVENTIONS:
Device: Wireless Physiologic Monitoring — YHE® BP Doctor Pro Blood Pressure Smartwatch, which is a commericially available device. The device can monitor heart rate, blood pressure and saturation.
  Arms: WIP

SUMMARY:
With over 18.5 million procedures performed worldwide and increasing, Cesarean section (CS) is the commonest surgical procedure. Inpatient monitoring is typically intense due to high risk for hemorrhage and other complications in the immediate post-operative period. Vital signs, including heart rate, blood pressure, saturation and temperature are monitored every 10-15 minutes. Maintaining this level of monitoring requires a significant dedication of human resources which is unattainable in resource-limited settings (RLS). Advancements in wireless physiologic monitoring offer a novel strategy to improve current monitoring levels. Through our project, we will evaluate the clinical use of a wireless physiological monitoring system for immediate postpartum monitoring in women after CS.

Our primary aims are:

I) To explore the clinical adequacy of wireless physiologic monitoring vs standard of care (SOC) monitoring immediately after uncomplicated Cesarean section in a RLS II) To explore the usability of wireless physiologic monitoring vs SOC monitoring among healthcare staff in a RLS

DETAILED DESCRIPTION:
Basic study design:

This pilot study will take place at Sir Ganga Ram Hospital, Lahore Pakistan as a cluster randomized clinical trial. Pakistan is a developing country with limited resources and a high maternal mortality rate of 189/100,000 live births. The tertiary hospital is located in the heart of historic city of Lahore which has a population of 11 million and the hospital has approximately 24,000 births per year. A conservative estimate of approximately 30 CS occur each day at the hospital.

Intervention:

Units will be randomized to the intervention, use of wireless physiologic monitoring system (WIP), or to SOC. The WIP system will be provided by YHE® BP Doctor Pro Blood Pressure Smartwatch, which is a commericially available device. The device can monitor heart rate

Randomization:

The hospital has 4 units and 1 operative theatre with post-operative ward. Each unit is responsible for all incoming operative cases on a rotating 1:1 randomization within each unit was not selected as there was a risk for contamination within each unit if healthcare staff realized that we were observing vital sign monitoring routines in the SOC arm.

Study population:

Peripartum women undergoing Cesarean birth. The target population is restricted to women undergoing CS due to the higher rates of morbidity and mortality compared to vaginal delivery.

Covariates:

We will extract relevant patient characteristics such as age, district of origin, education level, occupation, referred from another facility, relevant obstetric history (parity, gestational age at birth, antenatal complications, reason for CS) and medical comorbidities (hypertension, cardiac, pulmonary disease etc.) using chart review completed with patient history (with need to ensure no missing data).

Outcome Measures:

Aim I primary outcome: Composite adequacy score (CAS), which will be a composite of registered measurements of HR, saturation and BP measured during the first 2 hours after birth. Each registered vital sign will give 1 point. According to SOC, heart rate, blood pressure, respiratory rate, saturation, and temperature are supposed to be 0, 20, 40, 60, 80, 100 and 120 mins. We will compare the number of measurements displayed using the WIP system to SOC (manual registration of vital signs) in women participating in the study. Aim II primary outcome, the system usability scale is a validated 10 question, quick and easy survey which will be administered to healthcare staff attending women in the post-operative ward to investigate their views of the usability of the technology (0-100 point scale). Higher scores indicate better effectiveness (ability of users to complete tasks using the system, and the quality of the output of tasks), efficiency (level of resources consumed in performing tasks) and satisfaction (subjective feeling).

Methodology Aim I: Over 4 weeks, we will include full-term pregnant women according to standard hospital protocols. After informed consent, the pregnant women from units participating in the intervention arm will be asked to wear the WIP biosensor for 2 hours directly after their CS. Data will automatically be transferred to a central monitor/mobile app which will allow for tracking of vital signs by healthcare staff which will already have access to the monitor/app. Confirmed data transmission to the central monitoring station will be assessed and monitoring will begin automatically. HR, saturation and BP will be measured every 20 minutes according to the protocol. In units in the SOC arm, vital signs in patients will be measured by healthcare staff according to standard protocols. These vital signs are traditionally monitored by pulse-oximetry for saturation, manual wrist palpation for HR, and BP monitor-cuff which are entered into patient electronic charts. Data from patient charts will be extracted daily.

Aim II:

After the monitoring session, 'usability' will be measured by asking the healthcare staff in both arms of the study to complete a brief questionnaire based on the System Usability Scale. This evaluation tool will be administered only to those healthcare staff responsible for post-operative monitoring of women after CS. A score of 0-100 will be calculated. The scale has been found to be both robust and reliable. More specifically, healthcare staff will be asked to assess how easy the WIP biosensor was to use and interpret; whether they liked interacting with the system, whether they would be willing to use it again in the future. Similarly questions will be asked for the SOC strategy as well.

Data analysis and statistics:

Descriptive statistics will be used to summarize participant characteristics, obstetric and medical comorbidities. We will compare these covariates in the WIP intervention and the SOC arms to elucidate any major differences in the characteristics of the two groups. If we find possible confounders, and considering that this is a small RCT, we will formally consider adjusting for possible confounders in our statistical analyses. Outcome variables such as CAS, system usability score, early breast-feeding and skin-to-skin contact will first be described for both arms using absolute counts and percentages. Monitoring with the WIP device will be deemed "adequate" if there was >=94% capture of the maternal HR, RR, temperature, saturation, and BP every 20 minutes and if the captured data is successfully transferred to the central monitor for review (CAS=6.4 points out of 7.0). Additionally, for CAS (main outcome), in case of missing data (i.e. if monitoring was stopped before 2 hours), data will be assumed to be missing at random and we will use imputation to account for missing values. This data will be reported both in the original and after-imputation format. We will use linear regression to compare the outcome variables (CAS and system usability score: continuous variables) to our predictor variables (WIP intervention vs SOC: dichotomous). As mentioned earlier, in case of differences between the two groups, we will adjust the linear regression model accordingly and report both crude and adjusted values. Adjusted values will be reported using multiple linear regression. Since this is a small RCT, we do not anticipate finding any effect modifiers and are therefore not planning to stratify our results.

Power analysis:

Using the two sample t-test, with mean difference in CAS of 2 points, standard deviation of 3, two-sided alpha of 0.05 and a power of 0.8, the sample size per study arm should be 68 (each arm=34). We anticipate 20% of women to decline participation and increasing the sample size to 41 women per arm. However, due to the large number of operations occurring at the hospital, we plan to recruit at least 100 patients, with 50 patients in each arm of the study.

ELIGIBILITY:
Inclusion Criteria:

1) age ≥18 years, 2) undergoing CS for singleton pregnancy, 3) willing to stay in postpartum unit for at least 24 hours, 4) willing to wear sensor during their time at the post-operative monitoring ward, 5) able to provide consent 6) ability to speak Urdu/Punjabi or English

Exclusion Criteria:

1) women with complicated CS (e.g. due to excessive perioperative bleeding), 2) women with immediate-emergency CS due to fetal or maternal disease, 3) no informed, written consent 4) unwilling to wear devices or participate in questionnaires, or 5) known infectious disease including but not limited to viral hepatitis, tuberculosis, or HIV.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Cesarean sections are an operation performed only on pregnant females.
Enrollment: 100 (Actual)
Dates: Start 2023-10-22 (Actual); Primary Completion 2024-01-31 (Actual); Study Completion 2025-08-15 (Estimated)

PRIMARY OUTCOMES:
Clinical Adequacy Score | 4 months
  Composite adequacy score (CAS), is a composite of registered measurements of HR, saturation and BP measured during the first 2 hours after birth. Each registered vital sign will give 1 point.

SECONDARY OUTCOMES:
System Usuability Scale index | 4 months
  System usability scale is a validated 10 question, quick and easy survey which will be administered to healthcare staff attending women in the post-operative ward to investigate their views of the usability of the technology (0-100 point scale). Higher scores indicate better effectiveness (ability of users to complete tasks using the system, and the quality of the output of tasks), efficiency (level of resources consumed in performing tasks) and satisfaction (subjective feeling).

CONTACTS AND LOCATIONS:
Locations (1):
- Sir Ganga Ram Hospital, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No